CLINICAL TRIAL: NCT07067099
Title: Use of Plasma With Neutralizing Autoantibodies to Type I Interferons in Patients With Severe Refractory Flare-up of Hidradenitis Suppurativa
Brief Title: Neutralizing Interferon Type 1 in Hidradenitis Suppurativa
Acronym: NIHS-I
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/871; 2024-A01035-42 (Other: ANSM)
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Plasma therapy; Neutralizing type-1 interferon autoantibodies
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with severe acute flare Hurley stage III HS (Experimental): These patients present with refractory severe HS (Hurley stage III) flare treated with a transfusion of plasma containing high titre anti-IFN-1 auto-Antibodies.
  Interventions: Biological: Plasma with neutralizing autoantibodies to Type I Interferons

INTERVENTIONS:
Biological: Plasma with neutralizing autoantibodies to Type I Interferons — Transfusion of one unit of plasma containing high titre anti-IFN-1 autoantibodies

SUMMARY:
The purpose of the study is to evaluate the safety and type 1 Interferon (IFN) neutralization in patients with refractory severe Hidradenitis Suppurativa (Hurley stage III) after transfusion of plasma containing high titer anti-IFN-1 autoantibodies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18
* Patients with Hidradenitis suppurativa (Hurley stages II-III)
* Disease affecting at least two distinct anatomical areas,
* Total count of abscesses (A) and inflammatory nodules (N) ≥ 3
* IHS4 score ≥ 11
* Treatment of pain with opioids (≥ 20 mg/day)
* Resistance to previous use (for at least 3 months) of systemic antibiotics and TNF inhibitors (infliximab or adalimumab) or anti-IL17 (secukinumab).
* Vaccinations against SARS-CoV-2 and influenza up to date (or able to be carried out prior to the study procedure)
* Women using an effective method of contraception
* Signed informed consent

Exclusion Criteria:

* Active viral infection: herpes, VZV, HIV, HBV, HCV
* Active bacterial infection requiring systemic antibiotics
* Known allergy to blood components/plasma proteins
* Poor myocardial function (increased risk of for transfusion-associated circulatory overload) (symptomatic left ventricular failure and ejection fraction < 40%)
* Pregnant women
* Subjects with no social security coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety of transfusion of plasma containing high titer anti-IFN-1 auto-Antibodies | within 28 days of infusion
  Two aspects are considered when assessing safety:
  * Immediate serious adverse events (SAEs) (within 24 hours of infusion) and,
  * Delayed SAEs (within 28 days of infusion). Adverse events are coded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE V5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France